CLINICAL TRIAL: NCT00742846
Title: Effects of Intra-articular Versus Subacromial Steroid Injections on Clinical Outcomes in Adhesive Capsulitis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No enrollment
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, April Armstrong, Associate Professor, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB #26378
Record Dates: First submitted 2008-08-26; First posted 2008-08-28 (Estimated); Last update posted 2015-02-27 (Estimated); Status verified 2015-02

CONDITIONS: Adhesive Capsulitis
Keywords: Adhesive Capsulitis; Subacromial injection; Intraarticular injection
MeSH Terms: conditions — Bursitis | interventions — Lidocaine; Triamcinolone Acetonide

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1 (Active Comparator): The patient receives intra-articular steroid and local anesthetic injection under fluoroscopy.
  Interventions: Drug: Lidocaine + Kenalog
- Group 2 (Active Comparator): The patient receives subacromial steroid and local anesthetic injection under fluoroscopy.
  Interventions: Drug: Lidocaine + Kenalog
- Group 3 (Active Comparator): The patient receives intra-articular local anesthetic injection under fluoroscopy.
  Interventions: Drug: Lidocaine
- Group 4 (Active Comparator): The patient receives subacromial local anesthetic injection under fluoroscopy.
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Drug: Lidocaine + Kenalog — 5ml 1% Lidocaine + 1ml 40mg Kenalog®-10 into the shoulder joint
  Intra-articular injection with local anesthetic and steroid
  Other Names: Kenalog; Lidocaine
  Arms: Group 1
Drug: Lidocaine + Kenalog — 5ml 1% Lidocaine + 1ml 40mg Kenalog-10 into the subacromial space
  Local anesthetic and steroid in to the subacromial space
  Other Names: Lidocaine; Kenalog
  Arms: Group 2
Drug: Lidocaine — 5ml 1% Lidocaine alone into the shoulder joint.
  intra-articular local anesthetic injection
  Arms: Group 3
Drug: Lidocaine — 5ml 1% Lidocaine alone into the subacromial space.
  subacromial local anesthetic injection
  Arms: Group 4

SUMMARY:
The primary objective is to compare the clinical outcomes of patients with a clinical diagnosis of Adhesive Capsulitis who receive intra-articular versus subacromial steroid injections.

The secondary objective is to verify that steroid injections in combination with physical therapy lead to more favorable outcomes than local anesthetic injections in combination with physical therapy.

DETAILED DESCRIPTION:
Current treatment for Adhesive Capsulitis involves physical therapy. Steroid injections have not been shown to be as effective alone without the physical therapy. However, there are multiple studies that document the benefit of adding a steroid injection to the physical therapy. After a review of the literature, there are studies that compare different dosages of intra-articular steroid injections,value and site of the injections, and accuracy of clinical injections. There are currently no studies that compare the results after intra-articular versus subacromial injections in combination with physical therapy. This study would help us determine if location of the injection is a major factor in regaining motion. If it is significantly important to be intra-articular with the steroid, than it may be important to send patients for fluoroscopic guided injections routinely rather than risk the chance of not being within the joint.

ELIGIBILITY:
Inclusion Criteria:

* Meet clinical diagnosis of primary Adhesive Capsulitis
* Restriction in abduction to less than 130 degrees
* 50% reduction in external rotation as compared with the contralateral side
* An intact rotator cuff
* Between 18-75 years of age

Exclusion Criteria:

* Previous shoulder capsular surgery
* History of steroid injection(s) into affected shoulder
* Inability to provide informed consent
* Iodinated contrast dye allergy
* Allergy to lidocaine
* Other suspected shoulder pathology (i.e., tumor, rotator cuff rupture. infection, arthritis)
* Known bleeding diathesis
* Cervical spine pathology
* History of trauma to the shoulder
* Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-08; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
The primary goal of this study is to document the return of shoulder motion and resolution of adhesive capsulitis after intra-articular versus subacromial steroid injections versus anesthetic injections in combination with physical therapy. | 6-8 months

CONTACTS AND LOCATIONS:
Overall Officials: April Armstrong, MD, Principal Investigator — Penn State College of Medicine, Penn State Milton S. Hershey Medical Center
Locations (1):
- Penn State College of Medicine, Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

REFERENCES:
- [Background] Alvado A, Pelissier J, Benaim C, Petiot S, Herisson C. [Physical therapy of frozen shoulder: literature review]. Ann Readapt Med Phys. 2001 Mar;44(2):59-71. doi: 10.1016/s0168-6054(00)00062-3. French. PMID 11587654
- [Background] Andrieu V, Dromer C, Fourcade D, Zabraniecki L, Ginesty E, Marc V, Railhac JJ, Fournie B. Adhesive capsulitis of the shoulder: therapeutic contribution of subacromial bursography. Rev Rhum Engl Ed. 1998 Dec;65(12):771-7. PMID 9923046
- [Background] Arslan S, Celiker R. Comparison of the efficacy of local corticosteroid injection and physical therapy for the treatment of adhesive capsulitis. Rheumatol Int. 2001 Sep;21(1):20-3. doi: 10.1007/s002960100127. PMID 11678298
- [Background] Bert J. Shoulder injections for subacromial bursitis. Minn Med. 1996 Sep;79(9):6. No abstract available. PMID 8854664
- [Background] Carette S, Moffet H, Tardif J, Bessette L, Morin F, Fremont P, Bykerk V, Thorne C, Bell M, Bensen W, Blanchette C. Intraarticular corticosteroids, supervised physiotherapy, or a combination of the two in the treatment of adhesive capsulitis of the shoulder: a placebo-controlled trial. Arthritis Rheum. 2003 Mar;48(3):829-38. doi: 10.1002/art.10954. PMID 12632439
- [Background] Chen MJ, Lew HL, Hsu TC, Tsai WC, Lin WC, Tang SF, Lee YC, Hsu RC, Chen CP. Ultrasound-guided shoulder injections in the treatment of subacromial bursitis. Am J Phys Med Rehabil. 2006 Jan;85(1):31-5. doi: 10.1097/01.phm.0000184158.85689.5e. PMID 16357546
- [Background] Dacre JE, Beeney N, Scott DL. Injections and physiotherapy for the painful stiff shoulder. Ann Rheum Dis. 1989 Apr;48(4):322-5. doi: 10.1136/ard.48.4.322. PMID 2712613
- [Background] Dias R, Cutts S, Massoud S. Frozen shoulder. BMJ. 2005 Dec 17;331(7530):1453-6. doi: 10.1136/bmj.331.7530.1453. PMID 16356983
- [Background] Fouquet B, Griffoul I, Borie MJ, Roger R, Bonnin B, Metivier JC, Pellieux S. [Adhesive capsulitis: evaluation of a treatment coupling capsular distension and intensive rehabilitation]. Ann Readapt Med Phys. 2006 Mar;49(2):68-74. doi: 10.1016/j.annrmp.2005.09.001. Epub 2005 Sep 27. French. PMID 16229920
- [Background] de Jong BA, Dahmen R, Hogeweg JA, Marti RK. Intra-articular triamcinolone acetonide injection in patients with capsulitis of the shoulder: a comparative study of two dose regimens. Clin Rehabil. 1998 Jun;12(3):211-5. doi: 10.1191/026921598673772420. PMID 9688036
- [Background] Hollingworth GR, Ellis RM, Hattersley TS. Comparison of injection techniques for shoulder pain: results of a double blind, randomised study. Br Med J (Clin Res Ed). 1983 Nov 5;287(6402):1339-41. doi: 10.1136/bmj.287.6402.1339. PMID 6416401
- [Background] Kivimaki J, Pohjolainen T. Manipulation under anesthesia for frozen shoulder with and without steroid injection. Arch Phys Med Rehabil. 2001 Sep;82(9):1188-90. doi: 10.1053/apmr.2001.24169. PMID 11552189
- [Background] Loyd JA, Loyd HM. Adhesive capsulitis of the shoulder: arthrographic diagnosis and treatment. South Med J. 1983 Jul;76(7):879-83. doi: 10.1097/00007611-198307000-00016. PMID 6867799
- [Background] Parlier-Cuau C, Champsaur P, Nizard R, Wybier M, Bacque MC, Laredo JD. Percutaneous treatments of painful shoulder. Radiol Clin North Am. 1998 May;36(3):589-96. doi: 10.1016/s0033-8389(05)70047-6. PMID 9597076
- [Background] Richardson AT. Ernest Fletcher Lecture. The painful shoulder. Proc R Soc Med. 1975 Nov;68(11):731-6. doi: 10.1177/003591577506801137. No abstract available. PMID 53845
- [Background] Rizk TE, Pinals RS, Talaiver AS. Corticosteroid injections in adhesive capsulitis: investigation of their value and site. Arch Phys Med Rehabil. 1991 Jan;72(1):20-2. PMID 1985618
- [Background] Ryans I, Montgomery A, Galway R, Kernohan WG, McKane R. A randomized controlled trial of intra-articular triamcinolone and/or physiotherapy in shoulder capsulitis. Rheumatology (Oxford). 2005 Apr;44(4):529-35. doi: 10.1093/rheumatology/keh535. Epub 2005 Jan 18. PMID 15657070
- [Background] Tallia AF, Cardone DA. Diagnostic and therapeutic injection of the shoulder region. Am Fam Physician. 2003 Mar 15;67(6):1271-8. PMID 12674455
- [Background] White, AET, Tuite, J.D. The accuracy and efficacy of shoulder injections in restrictive capsulitis. Journal of Orthopaedic Rheumatology 1996; 9: 37-40.